CLINICAL TRIAL: NCT04273854
Title: Physician Optimised Post-partum Hypertension Treatment Trial
Acronym: POP-HT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 273353; FS/19/7/34148 (Other Grant/Funding Number: Funder: British Heart Foundation)
Record Dates: First submitted 2020-01-29; First posted 2020-02-18 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Pre-Eclampsia; Gestational Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All downstream data analysis will be done by investigators blinded to the allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will consist of physician-optimised self-management of post-partum BP. Women will follow a 'smartphone' app based algorithm for medication-titration, which will provide individualised dose titration advice.
  Interventions: Device: OMRON Evolv® blood pressure monitor (Blue-tooth® enabled) & Proprietary Smartphone POP-HT app®
- Control (No Intervention): The control arm will be managed as per usual NHS led care with assessment by their own health care professionals and adjustment of their medications as is needed. The BP of this group will be monitored and recorded at the same time-points and in the same manner as the intervention arm as will all other secondary outcome measures.

INTERVENTIONS:
Device: OMRON Evolv® blood pressure monitor (Blue-tooth® enabled) & Proprietary Smartphone POP-HT app® — The intervention will consist of physician-optimised self-management of post-partum BP. Women will follow a 'smartphone' app based algorithm for medication-titration, which will provide individualised dose titration advice. This is overseen and any change is approved by physicians who can review the uploaded readings and respond to tele-monitored abnormal readings in a timely fashion.
  Arms: Intervention

SUMMARY:
It has been shown in a pilot randomised controlled study [SNAP-HT [4]; REC 14/SC/1316] that blood pressure self-management during the post-partum period after hypertensive pregnancies, results in lower blood pressure after six months; even when medication has been stopped. The team now want to assess whether this blood pressure reduction can be reproduced in a larger, randomised, study (data analysis blinded) and whether the blood pressure lowering has additional benefits in terms of other cardiovascular and cerebrovascular changes known to occur in women who have had a hypertensive pregnancy. The investigators therefore plan to run a trial of self-management in the post-partum period, using updated Blue-tooth® enabled blood pressure monitoring coupled to physician-assisted dose titration to further advance the self-management aspect of the intervention. The physicians will be specialist clinicians who form part of the research team. The investigators will measure additional structural and functional end organ differences, using magnetic resonance imaging of the brain and heart as well as echocardiography and retinal imaging. This will provide insight into the impact of post-partum blood pressure control on the maternal cardiovascular system and how this associates with blood pressure changes. Together, these studies will help refine future intervention strategies in this cohort of patients.

DETAILED DESCRIPTION:
Summary of the Design ---------------------- The trial is a single centre, single blinded (the investigators will be unaware of which group the participants are allocated to), and randomised controlled study i.e. the group participants are put is allocated by chance. The study focuses on women who develop hypertensive disorders of pregnancy, which require ongoing treatment for blood pressure after birth at the time of discharge. These women will be randomised to one of two treatment arms: either usual care by GP/mid-wife/other NHS providers, or self -management of blood pressure. Women will be recruited from the John Radcliffe Hospital and this study will investigate the effectiveness of post-partum physician assisted self-management of blood pressure vs standard care over the first 6 (up to 9) months post-partum.

Trial Setting and participant profile

------------------------------------ The investigators aim to recruit 200 participants, of which 100 will be randomised to the intervention arm and 100 to the control arm. The intervention arm will comprise tele-monitored (remote) home blood pressure monitoring (including periods of home 24hr blood pressure monitoring) coupled to doctors overseeing medication self-management remotely. The control arm will receive 'standard' levels of NHS care from their GP and midwives and health visitors. All participants will be recruited from the Oxford Women's Centre at the John Radcliffe Hospital, which sees approximately 25 patients per month with hypertensive pregnancies (demonstrated in a local audit).

Trial participants --------------------- All participants will be females of childbearing age >18 years of age. Inclusion in the trial will require a clinician confirmed diagnosis of either gestational hypertension or pre-eclampsia as defined by NICE's latest guideline for this condition (NG 133), and the women must still require anti-hypertensive medication to control their blood pressure at the time of planned discharge.

Summary of the study visits

-------------------------- A flow chart of the proposed study visits can be seen in the protocol in section 9.7 and in appendix A of the protocol, which illustrates more clearly this textual description . The expected duration of participant involvement will be 6 (up to 9) months from enrolment to study completion and participants will be asked to attend four study visits after their pre-screening and enrolment: baseline, at 1 week, at 6 weeks and at 6-9 months. Although this study will only involve the four visits described above (outlined in appendix A) currently, further contact may be planned over the next 10 years to allow longitudinal follow up of this cohort. Details of the follow-up visits will be defined closer to the time and REC approval will be sought for any amendment/extension to this study to allow future contact. Additional consent will be sought from the participants to ensure they are happy to continue taking part.

Details of the study visits and procedures:

----------------------------------------- Both groups receive the same number of study visits, 4 visits for all participants.

Visit 1 (90 minutes) will take place in the first days after giving birth whilst participants remain on the post-natal ward in the Women's centre. The team will measure blood pressure, take some simple measurements e.g. weight, waist and hip circumference and scan their hearts (using ultra-sound just like they had of their babies). The team will then review the medical notes and blood tests and provide a questionnaire about lifestyle and diet, which can be completed later to shorten the visit. At the end of visit 1 participants will either be allocated to the intervention group or the control group. If allocated to the intervention group a separate member of the team will come and provide the participant with the blood pressure monitor (an OMRON EVOLV®) used for home monitoring. This team member will register and install the app on the participant's smartphone/tablet and teach the participant how to use it. They will therefore have plenty of time to practice with it whilst still in hospital.

Visits 2 and 3 (30 minutes) take place at weeks 1 and 6 weeks after discharge respectively and are to measure blood pressure, take some simple measurements e.g. waist, left arm and hip circumference, and to complete a brief questionnaire. These will be offered as a home visit, or as a visit to the Cardiovascular Clinical Research Facility (CCRF) at the John Radcliffe Hospital, depending on the women's preference, although based on prior experience it is expected most women will opt for home visits at this busy time in their lives. At the end of Visit 3 (week 6) there will be a 24 hour blood pressure monitor fitted, programmed to be silent to minimise disruption to the mum and the baby and the women will be provided with a stamped, addressed envelopes to post it back to CCRF. At the end of this visit, the team will run through the additional PIS relevant to the 4th visit again. This will allow participants to ask any questions about the longer final study visit up at the hospital, as the investigators are aware there is a lot to take in on the PIS and additional information sheet at the time of enrolment. The team will also call to discuss any further questions and plan child care for this longer visit in advance a few weeks prior to the 4th visit described below.

At 6-9 months there will be a slightly longer visit to CCRF in the John Radcliffe Hospital. Visit 4 (up to 4 hours) will involve measuring blood pressure again, doing another scan of the heart by ultra-sound, doing an MRI (magnet scan) of the heart and brain, and taking a blood test. There will also be a few other simple tests (not absolutely mandatory) but which are more exploratory secondary outcome measures for the study. These include: taking photos of the blood vessels in the back of the eye (retinal imaging, like an optician does), and doing some gentle exercise on a bike (akin to walking up a hill at a fast pace) during which the heart will be scanned to assess its response to exercise.

Each procedure that a participant will be asked to undergo during this study is summarised below in a little more detail: 1. Bed-side blood pressure measurement (10 minutes) Three blood pressure readings will be taken at intervals of 1 minute from the left arm using an automated blood pressure monitor (unless medical reason means the left arm cannot be used). This will require sitting at rest for 5 minutes prior to doing any measurements.

2. Echocardiogram scan (15 minutes) The team will perform an ultrasound (echocardiogram/echo) of the heart. This is a safe and painless procedure that takes 15 minutes. The Participant will be asked to lie on a couch on theirleft side. A probe is placed on the chest and lubricating jelly is used so the probe makes good contact with the skin. Ultrasound waves then create images of the heart on the scanner monitor. A female sonographer/scanner will be provided wherever possible and if not available, a female chaperone will be provided.

3. Vicorder® (Vascular Measures and Central Blood Pressures, 10 minutes): This involves lying flat on a cough and having two blood pressure cuffs fitted, one to the right arm and one around the right thigh. These are inflated and deflated three times at short intervals to acquire the readings. It is completely safe and painless.

4. Lifestyle and physical activity questionnaire (25 minutes): The questionnaire combines validated questionnaires taken from previous studies. Information will be collected on factors that affect blood pressure including: smoking frequency, alcohol and salt intake, exercise and family history. Questionnaires can be completed either during a study visit or at a later date and posted back to the study team (prepaid envelopes will be provided).

5. EQ-5D-5L Quality of Life questionnaire (5 minutes): Participants will be provided with an EQ-5D-5L questionnaire, which is a widely used and validated way of assessing quality of life at a set time-point. A trained study investigator will run through the structured questionnaire during the visit with the participant.

6. MRI Heart and Brain (1 hour including break) The MRI scanner is shaped like a polo mint, the hole inside measuring about 60 centimetres wide. MRI is safe and non-invasive and does not involve any ionising radiation (x-rays). However, because they use a large magnet to work, MRI scans are not suitable for everybody. Because of this, participants will be asked pre-screening safety questions to help determine if participants are able to take part. More detail about the MRI scan is provided on the additional information sheet given to participants before the 4th study visit. This additional information sheet also provides more detail about the optional sub-study of having gadolinium given (a commonly used contrast drug for MRI) to acquire an extra few images in those women who are no longer breast-feeding at that time-point. Additional consent will be sought and obtained for this sub-study prior to the MRI scan being performed.

7. Blood sampling (10 minutes) Blood samples will be collected (about 5 tablespoons (25mls) of blood). More detail is contained in the additional participant additional information sheet.

8. Fitting of a home blood pressure monitor (5 minutes, to be worn for 24 hours) and activity monitor (5 minutes, to be worn for 7 days and nights) The monitor consists of a blood pressure cuff, which will be fitted on the left arm (right if a specific medical reason precludes use of the left). A small bag will also be provided that is worn around the waist or shoulders, in which the blood pressure monitor is placed. Participants will be shown how to re-attach the monitor e.g. after a bath or shower or should it fall off. The BP monitor will automatically inflate hourly during the day and every other hour at night to minimise inconvenience at this busy time in their lives. Participants will be asked to wear the blood pressure monitor for 24 hours and to keep a brief blood pressure monitoring diary and information sheet to detail time participants went to sleep/awoke and any periods of cardiovascular activity such as running for the bus/cycling to work. A stamped addressed envelope will be provided to return the device after use. The activity monitor is waterproof and shock-proof and will be worn continually on the wrist for one week and again a stamped addressed envelope will be provided to return the device after use.

9. Retinal imaging (10 minutes) Photos will be taken of the back of the eyes just like at an optician. More information about this is provided on the additional PIS for the 4th study visit. To help keep personal information confidential, images will be 'de-identified' and assigned a study code. However, retinal images are unique so they can never be completely anonymous.

10. Cardiopulmonary Exercise Testing (CPET) with exercise echo (30 minutes) This involves gentle cycling on a stationary bicycle and doing a short ultrasound (echocardiogram) of the heart whilst exercising. There will be real-time measurement of heart rate and blood pressure. More information about this is provided on the Additional PIS.

11. Laser Speckle Tracking/Iontophoresis (15 minutes): this is an optional measure investigators will offer to 24 participants in each group of the trial. This will take an additional 15 minutes and is done twice; once at the baseline and once at the final/4th study visit in the 48 who agree. Participants will be asked to refrain from consuming caffeine (coffee, soft drinks, chocolate, etc.) for 4 hours prior to the forearm blood flow measurements. In this portion of the study, participants lay still in a bed. Two probes will be attached to the inner surface of the forearm. A special camera will be used to visualise blood flow in the skin of the forearm, which involves shining a red light on the skin. The investigators will use the probes to apply harmless solutions to the skin, while measuring the changes in the blood flow with the red light. This procedure causes no pain or discomfort.

The Intervention itself

------------------------- This next section only applies to participants in the intervention group and an additional intervention group information sheet will be provided for the participants allocated/randomised to this group in a written paper document as well as the information being available on the app and the study website. Women in this group will be asked to start measuring their blood pressure on the day of discharge from hospital using the OMRON EVOLV® monitor provided. This will mean taking 2 readings, 1 minute apart every morning after discharge. They will be asked to do this every morning, until they have had 5 consecutive days with blood pressure readings in the normal range (off medication). It is anticipated this will take 2-3 weeks following discharge based on our experience in our pilot study [SNAP-HT; REC 14/SC/1316].

After measuring the blood pressure, they will open up the POP-HT app on their smartphone/tablet, confirm it was them that took the blood pressure readings and click 'SYNC'. The app will then 'synchronise' with the OMRON EVOLV® monitor to upload the reading to the app and the secure study website hosted on the hospital's secure intranet (not the internet).

The smartphone/tablet will notify the participant if the readings are too high, too low or in the normal range. If they are high or low the app will ask them to repeat one more reading. If the reading is still high or low then the app will notify the participant and the specialist study doctors. The participant can then opt to receive a call from the study doctors to help adjust their own medication or they can choose see their own GP/mid-wife (further detailed information about this is available in the self-management information sheet).

Once a participant has 5 days in a row with readings in the normal range (off medication) they will be sent a notification/message reading "Thank you. Your blood pressure readings have all been normal since stopping treatment. Please change to once weekly readings for the remainder of the study." This will be until 6 months after the delivery of their baby/babies. The reason for the longer period of weekly monitoring is to ensure they do not have a late rise in your blood-pressure readings that requires further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Female, aged 18 years or above.
* Clinician confirmed diagnosis of either gestational hypertension or pre-eclampsia defined by NICE NG 133
* Requiring anti-hypertensive medication at the point of discharge from secondary care.
* Participant has clinically acceptable laboratory results and clinical course post-partum with no other adverse complicating factor requiring prolonged admission post-partum that would make participation unfeasible as judged by the CI. Examples would include stroke sequalae, ongoing DIC, the baby/babies requiring prolonged NICU/SCBU admission of >1 week.
* In the Investigator's opinion, is able and willing to comply with all trial requirements including ownership of a 'Smart-phone/Tablet' and willing to use the smart-phone app if randomised to that arm.
* Sufficient competence in English Language to follow the app instructions and partake in the study, as judged by the CI

Exclusion Criteria:

* Significant renal or hepatic impairment that would affect safe medication titration and adjustment as part of the trial, as deemed by the Investigator.
* Scheduled elective surgery (excluding caesarean sections) or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months.
* Any other significant disease or disorder, which, in the opinion of the Investigator, may either, put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* An absolute contra-indication to MRI (as per MRI safety questionnaire)
* Women with pre-existing hypertension will be excluded, as this is a separate pathology that would affect the efficacy of the study intervention and affect the primary and secondary outcomes of the study.

Additional exclusion criteria specific to the Gadolinium sub-study are:

* Breast feeding,
* eGFR <30ml/minute.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be female anatomy and genetically and have conceived and given birth
Enrollment: 200 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Diastolic Blood pressure (BP) | 6 months post-partum
  24 hour average diastolic BP measured by 24 hour ambulatory BP monitoring (ABPM)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordhsire
  - Cardiovascular Clinical Research Facility, Dept of Cardiovascular Medicine, University of Oxford, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No
Data will be made available, under certain circumstances, following data lock upon request to the study PI.

REFERENCES:
- [Derived] Lapidaire W, Kitt J, Krasner S, Bateman PA, Cutler HR, Barr L, Frost A, Tucker K, Suriano K, Kenworthy Y, Milner G, Lacharie M, Mills R, Roman C, Mackillop L, Aye C, Cairns A, Thilaganathan B, Chappell LC, Lewandowski AJ, McManus RJ, Leeson P. Brain Volumes After Hypertensive Pregnancy and Postpartum Blood Pressure Management: A POP-HT Randomized Clinical Trial Imaging Substudy. JAMA Neurol. 2026 Jan 5:e255145. doi: 10.1001/jamaneurol.2025.5145. Online ahead of print. PMID 41490362
- [Derived] Kitt J, Biasiolli L, Krasner S, Bateman PA, Cutler HR, Barr LC, Frost A, Tucker KL, Suriano K, Kenworthy Y, Lapidaire W, Lacharie M, Mills R, Roman C, Mackillop L, Aye CYL, Cairns AE, Thilaganathan B, Chappell LC, Lewandowski AJ, McManus RJ, Leeson P. Impact of Blood Pressure Self-Management on Vascular Remodeling After Hypertensive Pregnancy. Hypertension. 2025 Nov;82(11):1938-1947. doi: 10.1161/HYPERTENSIONAHA.125.24854. Epub 2025 Sep 4. PMID 40905148
- [Derived] Cutler HR, Kitt J, Sattwika PD, Finnigan LEM, Estevez-Fernandez A, Kenworthy Y, Suriano K, Frost A, Krasner S, Johnson C, McCourt A, Mills R, Tucker K, Cairns A, Roman C, Aye C, Mackillop L, Thilaganathan B, Chappell LC, Raman B, Lewandowski AJ, Lapidaire W, Leeson P. Subclinical Postpartum Renal Structure After Hypertensive Pregnancy Disorders. Hypertension. 2025 Nov;82(11):1948-1958. doi: 10.1161/HYPERTENSIONAHA.125.25130. Epub 2025 Aug 31. PMID 40886083
- [Derived] Kitt J, Fox R, Frost A, Shanyinde M, Tucker K, Bateman PA, Suriano K, Kenworthy Y, McCourt A, Woodward W, Lapidaire W, Lacharie M, Santos M, Roman C, Mackillop L, Delles C, Thilaganathan B, Chappell LC, Lewandowski AJ, McManus RJ, Leeson P. Long-Term Blood Pressure Control After Hypertensive Pregnancy Following Physician-Optimized Self-Management: The POP-HT Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1991-1999. doi: 10.1001/jama.2023.21523. PMID 37950919
- [Derived] Kitt J, Krasner S, Barr L, Frost A, Tucker K, Bateman PA, Suriano K, Kenworthy Y, Lapidaire W, Lacharie M, Mills R, Roman C, Mackillop L, Cairns A, Aye C, Ferreira V, Piechnik S, Lukaschuk E, Thilaganathan B, Chappell LC, Lewandowski AJ, McManus RJ, Leeson P. Cardiac Remodeling After Hypertensive Pregnancy Following Physician-Optimized Blood Pressure Self-Management: The POP-HT Randomized Clinical Trial Imaging Substudy. Circulation. 2024 Feb 13;149(7):529-541. doi: 10.1161/CIRCULATIONAHA.123.067597. Epub 2023 Nov 11. PMID 37950907
- [Derived] Kitt J, Frost A, Mollison J, Tucker KL, Suriano K, Kenworthy Y, McCourt A, Woodward W, Tan C, Lapidaire W, Mills R, Lacharie M, Tunnicliffe EM, Raman B, Santos M, Roman C, Hanssen H, Mackillop L, Cairns A, Thilaganathan B, Chappell L, Aye C, Lewandowski AJ, McManus RJ, Leeson P. Postpartum blood pressure self-management following hypertensive pregnancy: protocol of the Physician Optimised Post-partum Hypertension Treatment (POP-HT) trial. BMJ Open. 2022 Feb 23;12(2):e051180. doi: 10.1136/bmjopen-2021-051180. PMID 35197335

DOCUMENTS (1):
  • Informed Consent Form (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT04273854/ICF_000.pdf